CLINICAL TRIAL: NCT05042336
Title: A Phase Ib/Ⅱ Clinical Study to Explore the Effectiveness and Safety of Camrelizumab/Lenvatinib Combined With TACE in Patients With Borderline Resectable Hepatocellular Carcinoma
Brief Title: The Effectiveness and Safety of Camrelizumab/Lenvatinib Combined With TACE in Patients With Borderline Resectable HCC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LQ-BLHCC-210412
Record Dates: First submitted 2021-08-25; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Carrelizumab Plus Lenvatinib Combined With TACE; Borderline Resectable Hepatocellular Carcinoma
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- camrelizumab/lenvatinib combined with TACE (Experimental): Phase Ib trial： Ib-A group [camrelizumab q3w group]: TACE d1, camrelizumab 200mg, d1, 22, 43; Lenvatinib d7-43; Surgery d50; Group Ib-B [camrelizumab q2w group]: TACE d1, camrelizumab 200mg, d1, 15, 29; Lenvatinib d7-43; Surgery d50.
  Phase II trial： The enrolled patients received camrelizumab/lenvatinib combined with TACE treatment (a relatively safer treatment plan based on phase Ib), and the first imaging efficacy evaluation was performed at 6-8 weeks to evaluate surgical resection
  Interventions: Drug: camrelizumab/lenvatinib combined with TACE

INTERVENTIONS:
Drug: camrelizumab/lenvatinib combined with TACE — Lenvatinib 4mg qd body weight≤60,8mg；body weight>60,12mg
  Camrelizumab 200mg q2w/q3w

SUMMARY:
The effectiveness and safety of carmelizumab/lenvatinib combined with TACE in patients with borderline resectable hepatocellular carcinoma remain unknown. This subject is an open, single-arm, randomized, single-center, and phase Ib/II study according to simon's two phase design. In the phase Ib trial, the groups of patients were divided according to the frequency of camrelizumab: camrelizumab (q3w) plus lenvatinib and TACE group, certolizumab (q2w) plus lenvatinib and TACE group. In the phase II trial, the enrolled patients received camrelizumab/lenvatinib combined with TACE treatment (a relatively safer treatment plan based on phase Ib), and the first imaging efficacy evaluation was performed at 6-8 weeks for evaluation of surgical resection. If surgical resection is not possible, it is necessary to evaluate whether to continue TACE treatment. Afterwards, the imaging efficacy evaluation (RECISTv1.1) will be carried out every 6-8 weeks to evaluate whether to operate and determine the best operation time. If surgery is possible, choose to continue the treatment with camrelizumab and/or TACE according to the patient's condition after the operation until the disease progresses or intolerable toxicity, and the drug should be discontinued up to 2 years. Imaging examinations will be performed every 2-3 months within six months after the operation, and imaging examinations will be performed every 3-6 months after six months. Safety is based on physical examination, laboratory examination, drug-related adverse events, surgery-related adverse events, and serious adverse events. To explore the effectiveness and safety of camrelizumab/lenvatinib combined with TACE in patients with borderline resectable hepatocellular carcinoma, and to screen the predictive indicators of the efficacy and safety of the combined regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old;
2. HCC patients who have been pathologically diagnosed or meet the clinical diagnostic criteria of the "Primary Liver Cancer Diagnosis and Treatment Regulations (2019 Edition)" issued by the National Health Commission of China.
3. Borderline resectable HCC patients [1. The diameter of a single tumor>10 cm; 2. The number of tumors was 2-3 and the maximum diameter of any lesion>3 cm; 3. The number of nodules≥4; 4. The number of liver segments>2 and still confined to the half liver; 5. The lesion invades large blood vessels or is less than 1 cm away from the large blood vessels; 6. Portal vein cancer thrombosis Cheng's classification I/II; 7. No extrahepatic metastases];
4. Estimated survival period ≥ 3 months;
5. ECOG PS score 0-1 points;
6. Grading of liver function: Child A;
7. Have not received any anti-tumor system therapy (including chemotherapy, targeted drugs, immune monitoring point inhibitors, etc.) and local treatments (including HAIC, TACE, radiofrequency ablation, PVE, TARE, radiotherapy, etc.);
8. The main organ functions are normal, and the laboratory examination results within 7 days before enrollment meet the following conditions: White blood cells (WBC) ≥ 2.5×10^9/L, neutrophils (ANC) ≥ 1.5×10^9/L, platelets (PLT) ≥ 75×10^9/L, hemoglobin (HGB) ≥ 90g/L (without blood transfusion within 7 days or EPO tolerance); total bilirubin (TBI) ≤1.5×upper limit of normal range (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5×ULN; albumin ≥ 30g/L (not allowed within 14 days Supplement albumin or branched-chain amino acids); INR ≤1.5×ULN; blood creatinine (Cr) ≤1.5×ULN; urine protein ≤1+;
9. The patient voluntarily participated and signed an informed consent form.

Exclusion Criteria:

1. A history of severe allergic reactions to chimeric, human or humanized antibodies, or fusion proteins.
2. Pregnant or breastfeeding women, men and women of childbearing age who are unwilling or unable to take effective contraceptive measures;
3. History of other malignant tumors in the past 5 years, except: malignant tumors that have been treated for the purpose of curing, and there is no known active disease for ≥5 years before the first administration, and the potential risk of recurrence is low; fully treated non-melanoma skin cancer or malignant freckle-like nevus without evidence of disease; Carcinoma in situ that has been adequately treated without evidence of disease;
4. Medium or more pleural and ascites with clinical symptoms;
5. Active bleeding or abnormal blood coagulation (PT>16s, APTT>43s, INR>1.5×ULN), have bleeding tendency or are receiving thrombolysis, anticoagulation or antiplatelet therapy;
6. People with hepatic encephalopathy;
7. A history of gastrointestinal bleeding in the past 6 months or a clear tendency to gastrointestinal bleeding, such as: known local active ulcer lesions, stool occult blood++ or higher cannot be included in the group; if persistent stool occult blood +, gastroscopy an examination;
8. Patients with severe gastric fundus esophageal varices and need interventional therapy;
9. Untreated active hepatitis B. (Note: Hepatitis B subjects who have received antiviral therapy for 4 weeks and have an HBV viral load of less than 100IU/ml may be allowed to participate in the study)
10. Active hepatitis C, that is, those who are anti-HCV positive or HCV-RNA positive and have abnormal liver function;
11. People who have a history of psychotropic substance abuse, cannot be quit or have a history of mental disorders;
12. Patients who have received solid organ transplantation or bone marrow transplantation, or have had an active autoimmune disease requiring systemic treatment within 2 years before the first administration;
13. Existence of immunodeficiency disease or HIV infection;
14. There has been objective evidence showing that there are past or present pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, and severe lung function damage;
15. Major surgery on the liver or other parts within 4 weeks before the first administration, or minor surgery (such as simple resection, tooth extraction, etc.) within 1 week before the first administration;
16. Received the vaccine within 30 days before the first administration;
17. Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 4 weeks before the first administration;
18. Those who have received other experimental drugs or experimental medical devices within 4 weeks before the first administration;
19. Any significant clinical and laboratory abnormalities that the investigator believes will affect safety evaluators, such as: active infections that require systemic treatment, uncontrollable diabetes, and hypertensive patients undergoing 2 or less antihypertensive treatments Failure to drop to the normal range after drug treatment (systolic blood pressure>140mmHg, diastolic blood pressure>90mmHg), myocardial infarction within 6 months, abnormal thyroid function (>NCI CTCAE v4.0 level 1 standard), etc.;
20. Researchers believe that they are not suitable for entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | through study completion, an average of 1 year
  in order to explore more safe regimen
MPR | through study completion, an average of 1 year
  Survival tumors remaining ≤50% during surgery

SECONDARY OUTCOMES:
pCR | through study completion, an average of 1 year
  Refers to the pathological examination of tumor surgical specimens after transformation treatment without residual infiltrating tumor cells.
ORR | 8 weeks
  The incidence of CR (complete remission), PR (partial remission) and SD (stable disease).

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China